CLINICAL TRIAL: NCT06790641
Title: Pathways to Perinatal Mental Health Equity
Acronym: Pathways
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Nancy Byatt, Principal Investigator, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00001751
Record Dates: First submitted 2025-01-10; First posted 2025-01-24 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Perinatal Anxiety; Perinatal Depression; Social Determinants of Health (SDOH); Peer Support; Obstetric Care; Substance Use Disorder (SUD); Perinatal Depression, Substance Use
Keywords: implementation strategies; obstetric care; perinatal mental health; perinatal anxiety; perinatal depression; perinatal mood disorders; qualitative study; focus groups; mixed methods; perinatal care; peer mentors; peer support; healthcare-community partnership
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Cluster randomized design. Interventions will be implemented at level of clinical settings and all patients at the setting will be eligible to receive intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthcare-Community Partnership approach (Active Comparator): The Healthcare-Community Partnership approach will include the PRISM model plus PSI Peer Support specialists.
  Interventions: Behavioral: Program in Support of Moms (PRISM); Behavioral: PSI Peer Support
- Healthcare system approach (Active Comparator): The Healthcare system approach will include the PRogram In Support of Moms (PRISM) model alone.
  Interventions: Behavioral: Program in Support of Moms (PRISM)

INTERVENTIONS:
Behavioral: Program in Support of Moms (PRISM) — Program in Support of Moms (PRISM): a practice-level intervention with implementation support that helps obstetric practices integrate mental health care for perinatal individuals. To help obstetric practices implement pathways for screening, assessment, and a stepped intervention response for mental health problems and social determinants of health. PRISM offers training in trauma informed and equitable care, technical assistance, and implementation and change management support.
Behavioral: PSI Peer Support — Postpartum Support International (PSI) Peer Support: a service administered by PSI that pairs perinatal individuals with a volunteer peer mentor who provides support, psychoeducation, behavioral activation, and navigation services, which includes planning, goal setting, and practical tools to manage parenting and mental health symptoms.
  Arms: Healthcare-Community Partnership approach

SUMMARY:
Mental health conditions occurring during pregnancy and up to one year postpartum (the perinatal period) occur in 1 in 5 perinatal individuals. To improve mental health care during the perinatal period, this study will implement and compare a health care model of improving mood and anxiety disorder care in practices with a health care-community partnership model. The study will include 32 perinatal care settings across the United States. Half of them will have the health care model, the other half will have the health care-community partnership model. The study is designed to answer the question, "Should states and healthcare systems put resources into a healthcare system approach or a healthcare-community partnership approach to mental health care?" The results of this study will help states and healthcare systems decide how to develop pathways for increasing access to mental health care for pregnant and postpartum individuals.

DETAILED DESCRIPTION:
Mental health conditions are now the leading cause of death during pregnancy and the postpartum period (the perinatal period) in the United States. One in five individuals who are pregnant or one year or less postpartum experience a mood or anxiety disorder. Despite these risks and the availability of evidence-based treatments for mood and anxiety disorders that occur during this time, most do not receive adequate treatment, if any at all. Gaps in care loom largest for individuals who are Black or African American, Hispanic or Latino, American Indian or Alaska Native, or Native Hawaiian or other Pacific Islander. Thus, it is recommended that, in order to detect and address perinatal mood and anxiety disorders and related social inequities, screening be implemented in both healthcare and community settings.

In response, the study team has developed approaches for addressing mood and anxiety disorders in both healthcare and community settings caring for pregnant and postpartum individuals. These programs have been adopted across the United States. The study's community partner, Postpartum Support International (PSI), developed a national Peer Support Program that pairs individuals in need of support with a trained volunteer who has also experienced and fully recovered from a perinatal mood and anxiety disorder.

The study's research partner, UMass Chan, developed:

* A statewide program that offers support to patients and their medical professionals to help them both address mental health during pregnancy and the postpartum period.
* A national network of similar statewide programs to coordinate their efforts across the United States.
* A comprehensive approach to help obstetric care settings address mental health concerns among their patients.

Despite the benefits of these programs, investigators have learned that none of them is sufficient to address mental health challenges on their own.

In response, investigators will conduct this study to examine what happens when healthcare- and community-based teams' partner to deliver care for perinatal mood and anxiety disorders.

One of the aims of the study is to test the effectiveness of the Healthcare-Community Partnership between PSI and UMass Chan. Thirty-two perinatal care settings (e.g., clinics, practices, and health centers providing care to pregnant and postpartum individuals) across the United States will implement either a 1) health system-focused approach or 2) healthcare-community partnership approach to mental health. In the health system-focused approach, perinatal care settings will integrate screening, assessment, and treatment of mood and anxiety disorders into prenatal and postpartum care. The Healthcare-Community Partnership approach will include the health system-focused approach and PSI Peer Support. Thus, all patients getting perinatal care at the 32 clinical sites will be offered the intervention. The study team will then look at patient charts to see if patients receive treatment and/or peer support and whether depression and anxiety symptoms improve. Researchers will also look at how well perinatal care settings implement mental health care such as screening for depression, anxiety and social determinants of health; how often they identify patient needs; and how often they help patients find services to address those needs. The study team will also conduct surveys to look at racial bias and discrimination and burnout among the perinatal care professionals and peer mentors who are delivering the approaches.

Another aim is to prepare to spread what the study team learns to other perinatal care settings. Having learned that even proven approaches sometimes need to be adapted to make them work in new settings with new groups of people, the study team will meet and talk with patients, perinatal care professionals, and peer mentors who participate in the study to learn about their experiences. The study's goal is to identify barriers and facilitators to using these approaches on a wider scale.

The researcher-community partnership is led by PSI, a community-based organization promoting mental health awareness, support, and treatment for pregnant and postpartum individuals worldwide, and UMass Chan Medical School. The team includes experts in their own lived experience, psychiatry, psychology, obstetrics, health equity, public health, advocacy, statistics, social work and health services research. The research team will also work with a network of programs across the United States that aim to increase access to mental health care for pregnant and postpartum individuals.

To amplify the voices of individuals central to the study, researchers will also partner with the study's three advisory councils. The first council includes individuals with lived experience of mental health challenges and oppression. The second council includes the professionals and providers serving these populations. The third council involves members of teams working to increase access to mental health care. The study team will meet with the advisory councils every other month to discuss its approaches, study procedures and findings.

ELIGIBILITY:
Inclusion Criteria for perinatal care setting team members:

* Be employed by a participating perinatal care setting in a clinical role (including as an obstetrician-gynecologist, midwife, nurse practitioner, a nurse, a navigator, or administrative staff member who implemented the respective intervention during the study period).
* Be 18 years of age or older
* Provide verbal consent prior to the focus group or interview
* Be proficient in English

Inclusion Criteria for peer mentors:

* Have completed PSI training to be a peer mentor
* Be 18 years of age or older
* Provide verbal consent prior to the focus group or interview
* Be proficient in English

Inclusion Criteria for perinatal individuals:

* Have received perinatal care at a study partnering perinatal care setting during the study period
* Be 18 years of age or older
* Provide verbal consent prior to the focus group or interview
* Be proficient in English or Spanish

Exclusion Criteria:

An individual who does not meet the inclusion criteria listed above will be excluded from participation in this study. There are no additional exclusion criteria.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1270 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2030-10-01 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in depression score as measured by either Edinburg Postnatal Depression Scale (EPDS) or Patient Health Questionnaire (PHQ9) | Baseline to up to 13 months postpartum
  Perinatal individual depressive symptoms will be determined from their medical charts, through the screening questionnaire used by their care setting. The screener may be the Edinburgh Postnatal Depression Scale (EPDS) or the Patient Health Questionnaire-9 (PHQ-9). The 10-item EPDS is the most widely used measure of perinatal depression symptoms. The 9-item PHQ-9 is the most widely-used measure of depression symptoms across the lifespan and the second most widely used measure during the perinatal period.
Proportion of perinatal individuals with evidence of initiation of treatment/support in their medical chart | Baseline to up to 13 months postpartum
  Perinatal individual initiation of treatment/support will be determined by their medical charts' indication that they have received treatment or support. Treatment or support is defined as one initial mental health assessment or treatment visit, peer support encounter, or currently on medication for depression or anxiety. Perinatal individuals will receive a score of 1 if they initiated treatment or support or a score of 0 if they did not initiate treatment or support. This outcome refers to the % of perinatal individuals who received treatment or support.

SECONDARY OUTCOMES:
Perinatal individual anxiety symptoms | Baseline to up to 13 months postpartum
  Perinatal individual anxiety symptoms will be determined from their medical charts, through results of the Generalized Anxiety Disorder Scale (GAD-7). The GAD-7 has seven items assessing anxiety severity and is validated in perinatal populations.

OTHER OUTCOMES:
Perinatal individual screening, assessment, treatment, and follow-up | Baseline to up to 13 months postpartum
  Whether perinatal individuals have received screening, assessment, treatment, and follow-up for mental health concerns will be determined from their medical charts. Receipt of screening and results (positive screen versus not) of screening will be determined from medical charts. Screeners will include Edinburgh Postpartum Depression Scale [EPDS], Nine-item Patient Health Questionnaire [PHQ-9], or Seven-item Generalized Anxiety Disorder scale [GAD-7]. Higher scores on these scales indicate higher symptom severity. Recognizing that a positive screen is not synonymous with a diagnosis, we will code mental health assessment (including administration and results of secondary screeners), as well as follow-up. Treatment follow-up will be defined as an average of ≥1 mental health service every month over 3 months or currently on medication for depression or anxiety during the study window.
Perinatal Individuals Social Determinants of Health (SDOH) screening and referral | Baseline to up to 13 months postpartum
  Perinatal Individuals' Social Determinants of Health (SDOH) screening and referral will be determined by review of their medical charts. Researchers will look for completion of the steps in the WE CARE process (screening, discussion with care professionals, and referral for unmet needs) and responses to the 12-item WE CARE screener.
Workforce capacity and support for engaging in mental health care | Baseline to up to 2 years post-implementation
  Perinatal care setting staff and peer mentor capacity and support for engaging in mental health care will be measured by the Pathways survey. To develop the Pathways survey, we carefully reviewed questions and constructs from the Mini-Z Single-Item Burnout Scale, the Trauma-Informed System Change Instrument questionnaire, the Kaiser Family Foundation's National Survey of Physicians, and the Determinants of Implementation Behavior Questionnaire. Rather than focus on participants' behaviors (for which we will collect data from electronic medical records and PSI administrative databases), the survey emphasizes questions on participants' perspectives regarding motivation and capacity to deliver mental health care, beliefs about consequences, and trust. Higher scores on the Pathways survey indicate higher capacity and support for engaging in mental health care.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Byatt, DO, MS, MBA, Principal Investigator — UMass Chan Medical School and UMass Memorial Health
Locations (1):
- UMass Chan Medical School, Shrewsbury, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No